CLINICAL TRIAL: NCT02619630
Title: Multicenter Study of Risk-adapted Treatment for T-lineage ALL of Young Adults (18-59 Years Old): Evaluating the Efficacy of a Nelarabine Based Consolidation and Maintenance in High-risk Patients
Brief Title: Multicenter Study of Risk-adapted Treatment for T-lineage ALL of Young Adults (18-59 Years Old)
Acronym: GRAALL-2014/T
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOM12629_2
Record Dates: First submitted 2015-11-25; First posted 2015-12-02 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-02

CONDITIONS: T-cell Adult Acute Lymphoblastic Leukemia
MeSH Terms: interventions — nelarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-Risk (HR) patients (Experimental): Nelarabine during consolidation and maintenance
  Interventions: Drug: nelarabine

INTERVENTIONS:
Drug: nelarabine — Nelarabine 1500 mg/m2/d (IV 2h) : D1, D3, D5 Cyclophosphamide 150 mg/m2/d (IV 3h) : D1, D3 etoposide (VP-16) 75 mg/m2/d (IV 1h) : D1, D3 granulocyte-colony stimulating factor 5 µg/kg/d (SC) : D7 until neutrophil >1 Giga/Liter
  for a maximum of 5 blocks

SUMMARY:
The purpose of this study is to evaluate the efficacy of nelarabine-based consolidation and maintenance therapy in term of relapse-free survival (RFS) in high-risk (HR) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Whose blood and bone marrow explorations have been completed before the steroids prephase
2. aged 18-59 years old with a not previously treated (including IT injection) T-ALL newly-diagnosed according to the WHO 2008 definition with > 20% bone marrow blasts
3. With Eastern Cooperative Oncology Group (ECOG) performance status < 3
4. With or without central nervous system (CNS) involvement or testis
5. Without other evolving cancer (except basal cell carcinoma of the skin and "in situ" carcinoma of the cervix) or its chemo or radio-therapy treatment finished at least since 6 months
6. Having signed a written informed consent
7. With efficient contraception for women of childbearing age (excluding estrogens and IUD)
8. Having received or being receiving steroid prephase
9. With health insurance coverage

Exclusion Criteria:

1. With lymphoblastic lymphoma and bone marrow blasts < 20%, Burkitt-type ALL or with antecedents of chronic myeloid leukemia (CML) or other myeloproliferative neoplasm
2. With contra-indication to anthracyclines or any other general or visceral contra-indication to intensive therapy except if considered related to the ALL:

   * Aspartate transaminase (AST) and/or alanine transaminase (ALT) > 5 x upper limit of normal range (ULN)
   * Total bilirubin ≥ 2.5 x upper limit of normal range (ULN)
   * Creatinine > 1.5 x upper limit of normal range (ULN) or creatinine clearance <50 mL/mn
3. Myocardial infarction within 6 months prior to inclusion in the trial, cardiomyopathy (NYHA grade III or IV), left ejection ventricle fraction (LEVF) < 50% and/or RF < 30%,
4. Active severe infection or known seropositivity for HIV or Human T cell leukemia/lymphoma virus type 1 (HTLV-1) or active hepatitis B or C
5. Other active malignancy
6. Pregnant (beta-Human Chorionic Gonadotropin (hCG) positive) or nursing woman
7. Women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least three months thereafter. Patients not willing to ensure not to beget a child during participation in the study and at least three months thereafter
8. Treated with any other investigational agent or participation in another trial within 30 days prior to entering this study
9. Not able to bear with the procedures or the frequency of visits planned in the trial
10. Unable to consent, under tutelage or curators, or judiciary safeguard

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 275 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 4 years

SECONDARY OUTCOMES:
Overall survival | 4 years
Cumulative incidence of relapse | 4 years
Non relapse mortality (NRM) | 4 years
Disease free survival censored at allograft in first complete remission (CR) | 4 years
Cumulative incidence of relapse censored at allograft in first complete remission (CR) | 4 years
Overall survival censored at allograft in first complete remission (CR) | 4 years
Non relapse mortality (NRM) censored at allograft in first complete remission (CR) | 4 years
Minimal residual disease (MRD) | within 1 year
Proportion of patients having received the 5 cycles of nelarabine | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology, Paris, France

REFERENCES:
- [Derived] Boissel N, Chevret S, Rigal-Huguet F, Leguay TT, Hunault M, Graux C, Chalandon Y, Delabesse E, Hicheri Y, Chevallier P, Balsat M, Pastoret C, Escoffre-Barbe M, Pasquier F, Joris M, Thiebaut A, Huynh A, Dhedin N, Lemasle E, Bonmati C, Maury S, Guillerm G, Berceanu A, Schanz U, Cluzeau T, Turlure P, Rousselot P, De Prijck B, Grardel N, Bene MC, Lafage-Pochitaloff M, Cuccuini W, Ifrah NH, Lheritier V, Asnafi V, Clappier E, Dombret H. Age-adapted chemotherapy and MRD-oriented transplant for Ph-negative acute lymphoblastic leukemia: the GRAALL-2014 trial. Blood. 2025 Oct 24:blood.2025029611. doi: 10.1182/blood.2025029611. Online ahead of print. PMID 41135009